CLINICAL TRIAL: NCT05694247
Title: A Single Arm, Open Label, Multicenter Clinical Investigation to Evaluate the Clinical Safety and Performance of the CorNeat Keratoprosthesis, for Treatment of Corneal Blindness
Brief Title: Study to Evaluate the Clinical Safety and Performance of the CorNeat KPro for Treatment of Corneal Blindness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CorNeat Vision Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS-35932
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-02

CONDITIONS: Corneal Disease; Corneal Opacity; Corneal Injuries
MeSH Terms: conditions — Corneal Diseases; Corneal Opacity; Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CorNeat KPro (Experimental): Intraocular implantation of the CorNeat KPro
  Interventions: Device: CorNeat KPro

INTERVENTIONS:
Device: CorNeat KPro — The optical component of the CorNeat KPro will be implanted into a circular disc of the cornea (as performed in standard penetrating keratoplasty surgery) and the skirt component will be embedded under a 360º conjunctival flap.

SUMMARY:
A Single Arm, Pivotal, Open Label, Multicenter Clinical Investigation to Evaluate the Clinical Safety and Performance of the CorNeat Keratoprosthesis, for Treatment of Corneal Blindness

DETAILED DESCRIPTION:
This clinical trial will assess the clinical safety and performance of the CorNeat Keratoprosthesis (KPro), a synthetic, artificial cornea for or the treatment of corneal blindness in subjects who are not candidates for traditional corneal transplant.

40 subjects who are willing to take part in the study will undergo screening examinations to verify their eligibility.

The CorNeat KPro will be implanted unilaterally in eligible subjects. Follow up procedures will be performed at 1 day, 1 week, 2 weeks, 1, 2, 3, 4, 5, 6,8, 10,12,15,18,21 and 24 months post-surgery and will include clinical assessment of the implanted eye using slit-lamp biomicroscopy, intra ocular pressure measurement and ocular imaging. Additionally, subjects' visual acuity will be assessed and recorded throughout the 24 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 21 and ≤ 80 years on the day of screening
2. Candidates must have the ability and willingness to attend all scheduled visits and comply with all study procedures
3. Legally blind (BCVA of 6/120 or worse in the better eye) in one or two eyes. In case of unilateral blindness - BCVA of Counting Fingers (CF) from 1 meter or worse in the operated eye
4. Keratoprosthesis surgery is indicated in cases when keratoplasty is not a reasonable option or following a verifiable history of prior failed corneal transplantation.
5. Indications that fall under poor candidate for keratoplasty include but are not limited to: herpetic keratitis, vascularized corneal scar, Ocular Cicatricial Pemphigoid, alkali burn, Steven Johnson Syndrome, and limbal stem cell deficiency;
6. Adequate tear film and lid function
7. Perception of light in all quadrants
8. Female patients of childbearing age must have negative pregnancy test at screening and agree to use an effective method of contraception throughout the study.

Exclusion Criteria:

1. Reasonable chance of success with traditional keratoplasty
2. Current retinal detachment
3. Connective tissue diseases or severely scarred conjunctiva in the target eye
4. End stage glaucoma or evidence of current uncontrolled glaucoma
5. History or evidence of severe inflammatory eye diseases (i.e. conjunctivitis, uveitis, retinitis, scleritis)
6. Active inflammation of the conjunctiva in one or both eyes
7. History of ocular or periocular malignancy
8. History of extensive keloid formation
9. Any known intolerance or hypersensitivity to topical anaesthetics, mydriatics, or component of the device
10. Ocular ischemic syndrome
11. Signs of current infection, including fever and current treatment with antibiotics
12. Severe generalized disease that results in a life expectancy shorter than two years
13. Any clinical evidence that the investigator feels would place the subject at increased risk with the placement of the device
14. Corneal thickness less than 400 or higher than 1,200 microns in any region of the pachymetry map of the eye intended to be operated
15. Currently pregnant or breastfeeding
16. Participation in any study involving an investigational drug or device within the past 30 days or 5 half-lives of the drug (whichever longer) or ongoing participation in a study with an investigational drug or device
17. Intraoperative complication that would preclude implantation of the study device
18. Hemoglobin A1C (HbA1c) higher than 8% at screening indicating unbalanced diabetes and/or target organ damage associated with diabetes
19. Patients requiring anticoagulation treatment, which cannot be interrupted for the surgical procedure
20. Vulnerable populations - minors, pregnant women, prisoners, sponsor or study institution employees, military persons, terminally ill, comatose, physically and intellectually challenged individuals, institutionalized patients and refugees
21. Subjects with corneal disorders located outside the central 7 mm, such as Mooren ulcer, peripheral ulcerative keratitis, and necrotizing herpetic keratitis (if located outside the central 7 mm of the cornea)
22. Patients with a functioning trabeculectomy or existing Microinvasive Glaucoma Surgery (MIGS) device that shunts aqueous from the anterior chamber into the subconjunctival space

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment | Throughout 24 months post-op
  The frequency of all Unanticipated Adverse Device-related Events (UADE) during and following implantation

SECONDARY OUTCOMES:
Retention rate | 24 months post-op
  The number of retained devices at the end of 24- months follow up period will be calculated
Change in Best Corrected Distance Visual Acuity (BCDVA) from baseline | Throughout 24 months post-op
  Visual acuity will be measured with ETDRS format charts. The number of patients with BCDVA better than 6/120 at 24 months after

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - UHN - University Health Network, Toronto, Ontario
- France (2):
  - CHU de Montpellier, Montpellier
  - Hopital Fondation Adolphe de Rothschild, Paris
- Rabin Medical Center - Beilinson, Petah Tikva, Israel
- Amsterdam UMC - Location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided